CLINICAL TRIAL: NCT04254302
Title: WECARE - Using Telerehabilitation to Support Families of Children With Motor Difficulties Aged 3-8 Years Old: A Patient-centred, Mixed-method Innovative Pragmatic Trial
Brief Title: Using Telerehabilitation to Support Families of Children With Motor Difficulties Aged 3-8 Years Old
Acronym: WeCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Chantal Camden, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-3429
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Motor Disorders
Keywords: Tele-intervention; Motor delay; Child; Parental support
MeSH Terms: conditions — Motor Disorders; Psychomotor Disorders

STUDY DESIGN:
Intervention Model Description: The family will be the unit of randomization. A web-based randomization service will allocate participants to either usual care or the WECARE intervention (1:1). To ensure equal distribution of participants between arms, permutated blocks of variable (2:4:6) size will be generated. No stratification or minimization strategies will be used. Participants will be invited to set their motor-performance goals before allocation to avoid the influence of the allocation group on goals selection.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded data collection specialists will conduct pre-intervention COPM and PEDI-CAT interviews, as well as post-intervention PEDI-CAT interviews. All other measures are self-completed online. The researchers and data analyst will also be blinded to participant allocation. Participants will be made aware of their allocation group following goals selection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants randomized into the control arm will receive usual care as per the service delivery models and pathways planned in their region. As a pragmatic trial, no attempt will be made to standardize practices which may vary across professionals. Usual practices may be categorised as either reference to online websites deemed appropriate by their healthcare professional, general recommendations, referral for services, or none of the above.
- Experimental (Experimental): WECARE intervention include: 1) 30-minute appointments with an occupational therapist or a physiotherapist, as part of a multidisciplinary team, to problem-solve the child's motor performance issues, provide recommendations to stimulate the child's motor development, and intervene online directly with the child, if needed; offered bimonthly during the first three months, then on a patient-identified needs-basis. 2) A chat function where participants can privately contact the therapist; flexible access as per participant needs. 3) A forum open to all intervention group participants where they can communicate with each other or with the therapist, who will also act as a forum moderator; flexible access as per participant needs. 4) Access to static online information via relevant websites and resources on child development; flexible access based on participant needs.
  Interventions: Other: WECARE web platform

INTERVENTIONS:
Other: WECARE web platform — The WECARE intervention allows families of children with motor difficulties to access rehabilitation therapists. The primary therapist will be an occupational therapist or a physiotherapist who will have one day a week to deliver the intervention. The therapist will act as case manager to connect families with community-based services available in their region and work, according to a transdisciplinary model, with an interdisciplinary team on a needs-based basis. Patient engagement with the therapists and in the WECARE intervention will be ensured by the collaborative coaching approach used by therapists to attain meaningful motor outcomes, as selected by the primary respondent.
  Arms: Experimental

SUMMARY:
Background: Many children (about 1 child out of 20) have motor delays that are sometimes seen as "minor" and are not immediately explained by a specific diagnosis. These children are often underserved by existing health and rehabilitation services even though they are at risk of developing important negative outcomes in the long run. The most recent scientific evidence indicates that motor delays can be effectively addressed via early interventions supporting families and stimulating the child's development. Some researchers have proposed that such interventions could be efficiently and conveniently delivered online but no patient-centred, interactive online intervention has been formally trialed in Canada for children with motor delay and their families.

Objectives: The goal of this study is to determine whether an online intervention can support families of children with motor delay. This study will determine whether the online intervention can improve the child's motor skills and parental self-efficacy, decrease parental stress, as well as increase the quality of life of both the parent and child.

Description: The investigators will recruit 118 families of children with motor delay, 3 to 8 years of age, who are not yet receiving public rehabilitation services. These children will have been identified as at-risk of motor difficulties by their parents who will have completed a self-reported screening test for motor difficulties. Families will be randomly assigned to one of two groups: 1) control group (usual care) or 2) intervention group (access to the WECARE web platform, including one-on-one virtual meetings with health professionals, group and private discussions, verified resources). This study, conducted in Quebec, will be led by researchers, telerehabilitation experts, decision makers and patient advocates.

Relevance: This study will evaluate an innovative, convenient and accessible intervention providing assistance for an important yet underserved population of children and their families.

DETAILED DESCRIPTION:
Detailed objectives:

The overarching goal of this patient-centred, mixed-methods, randomized, innovative pragmatic trial is to evaluate the effectiveness of the WECARE intervention for children aged 3-8 years with motor difficulties living in Quebec. The primary objective is to evaluate, in comparison to usual care management, the effectiveness of the WECARE program for improving the child's performance on parent-identified motor functioning targets. Secondary objective is to evaluate the effect of the intervention on children's functioning, parental self-efficacy, parental stress, as well as the quality of life of both the parent and child.

Detailed design: A patient-centred innovative pragmatic randomized controlled trial documenting real-world effectiveness of the WECARE intervention, offered to families of children with motor difficulties living in Quebec and receiving no public rehabilitation services. A primary respondent (i.e., parent or legal guardian) will be identified but the whole family will have access to the WECARE intervention.

This trial was designed according to the latest guidelines on pragmatic trials, using the gold-standard CONSORT guidelines, and the TElehealth in CHronic Disease (TECH) conceptual framework.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child aged 3-8 years old at risk of motor difficulties, as confirmed via the DCD-Questionnaire or Little DCD-Q
* Have at least one motor-related COPM objective at T0
* Live in Quebec.

Exclusion Criteria:

* Children receiving public rehabilitation services for their motor difficulties at time of enrolment (i.e. receiving either physiotherapy or occupational therapy services)
* Families whose parents could not provide a single motor performance related goal to inform the intervention.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Structured interview and numerical rating scales : before intervention. Numerical rating scales only : every 3 months for 12 months (i.e 3 months, 6 months, 9 months and one year after the beggining of the intervention)).
  The COPM uses a structured interview to identify intervention goals. Ten-point numerical rating scales are then used to identify importance, actual performance and satisfaction with performance for each selected goal. Higher scores indicate higher importance, better performance and higher satisfaction with the child's performance. An increase of more than 2 points on the 10-point numerical rating scale is considered as a meaningful clinical difference and will be used as an indication of the attainment of the child's motor performance goal. The COPM does not require any physical or hands-on materials, which is consistent with an online trial.

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory - computer adaptive test (PEDI-CAT) | Baseline and 1 year after the beggining of the intervention (pre- and post-intervention]
  The PEDI-CAT is a parent-reported adaptative questionnaire for parents of children between the ages of 0 and 20 years old. Each question is selected by the computer algorithm based on the child's socio-demographic data and answers to previous questions. A maximum of 15 questions are asked for each domain. The number of items needed to establish the child's score may vary according to the stopping rules of the algorithm. For each question, parents indicate their child's ability to participate in a presented activity (e.g. Putting on socks) on a 4-points scale ranging from "Unable = Can't do, doesn't know how or is too young" to "Easy = Does with no help, extra time, or effort, or child's skills are past this level". The score for each subscale is expressed in T-scores. The Daily activities and Mobility subscales of the Short Form PEDI-CAT will be used in this project.
Parental Knowledge and Skills Questionnaire (PKSQ) | Baseline and 1 year after the beggining of the intervention (pre- and post-intervention]
  The PKSQ has been validated to evaluate the self-efficacy of parents of children with Developmental coordination disorder (DCD) aged 0-18 years-old. An adapted version of the PKSQ will be used to remove the focus from DCD and ensure its relevance for all motor difficulties. The adapted PKSQ includes two out of the three constructs of the original version of the PKSQ. The adapted version includes 14 questions about parental understanding of motor difficulties and their perception of their capacity to manage their child's motor difficulties. Questions are scored by the parent on a 7-point Likert scale ranging from "Not at all" to "To a very great extent".
Parental Stress Scale (PSS) | Baseline and 1 year after the beggining of the intervention (pre- and post-intervention]
  Parental stress will be measured with the Parental stress scale (PSS). The PSS includes 18 questions about parental feelings and experience of parenting. Each statement is scored on a 5-point Likert scale (1=Strongly agree to 5=Strongly disagree). Higher scores indicate lower parental stress.
Six Dimension Short-Form Health Survey (SF-6D) | Baseline and 1 year after the beggining of the intervention (pre- and post-intervention]
  Changes in the parent's quality of life will be measured with the Six Dimension Short-Form Health Survey (SF-6D). The SF-6D is a tool measuring health utilities in adults. It includes items on physical and social functioning, role limitations, pain, mental health and vitality. The total score is reported on a scale ranging from 0,29 to 1, where 1 represents a perfect health (i.e. a greater score means a better health).
Health-Related Quality of Life Utility Measure for Pre-School Children (HuPS) | Baseline and 1 year after the beggining of the intervention (pre- and post-intervention]
  Changes in children's quality of life will be measured with the Health-Related Quality of Life Utility Measure for Pre-School Children (HuPS) tool. The HuPS includes 12 questions about the child's abilities rated on a 3- to 5-point scale (e.g.: seeing, speaking, using hand and fingers, selfcare). Changes in the parent's quality of life will be measured with the Six Dimension Short-Form Health Survey (SF-6D). The SF-6D is a tool measuring health utilities in adults. It includes items on physical and social functioning, role limitations, pain, mental health and vitality. The total score is reported on a scale ranging from 0 to 1, where 1 represents a perfect health (i.e. a greater score means a better health).

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Camden, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No